CLINICAL TRIAL: NCT04420871
Title: Pharmacokinetic and Safety Comparison of Two Capecitabine Tablets in Patients With Colorectal or Breast Cancer Under Fed Conditions: a Multicenter, Randomized, Open-label, Three-period, and Reference-replicated Crossover Study
Brief Title: Pharmacokinetic and Safety Comparison of Two Capecitabine Tablets in Patients With Colorectal or Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-KPTB-150
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Patient Participation
Keywords: Capecitabine; Bioequivalence; Pharmacokinetics
MeSH Terms: conditions — Patient Participation | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, open-label, three-period, and reference-replicated crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- capecitabine reference formulation at a single dose of 150 mg (Active Comparator): 150 mg of Xeloda® produced by Genentech USA, Inc., a subsidiary of the company, was used as the reference intervention in this study.
  Interventions: Drug: 150 mg of Xeloda®
- capecitabine test formulation at a single dose of 150 mg (Experimental): The tablet of 150 mg of capecitabine from Qilu Pharmaceutical Co., Ltd. (17H0053DE4, Jinan, Shandong Province, China) was used as the test formulation.
  Interventions: Drug: 150 mg of capecitabine

INTERVENTIONS:
Drug: 150 mg of Xeloda® — Subjects were allocated to one of three groups randomly and equally with a 1-day wash time period. 150 mg of Xeloda® produced by Genentech USA, Inc., a subsidiary of the company, was used as the reference intervention in this study.The subjects randomly received single oral administration of 150 mg of Xeloda®.
  Arms: capecitabine reference formulation at a single dose of 150 mg
Drug: 150 mg of capecitabine — Subjects were allocated to one of three groups randomly and equally with a 1-day wash time period.The tablet of 150 mg of capecitabine from Qilu Pharmaceutical Co., Ltd. (17H0053DE4, Jinan, Shandong Province, China) was used as the test formulation.The subjects randomly received single oral administration of 150 mg of capecitabine.
  Arms: capecitabine test formulation at a single dose of 150 mg

SUMMARY:
A multicenter, randomized, open-label, three-period, and reference-replicated crossover study was conducted in 48 patients with colorectal or breast cancer under fed conditions to assess the bioequivalence between two formulations of capecitabine.

DETAILED DESCRIPTION:
This was a multicenter, open, random, balanced, three-period, three-sequence and semi-repetitive cross study with 48 subjects. Eligible subjects were randomly assigned in a 1:1:1 ratio to receive one period of test formulation or two period of reference formulation, followed by a 1-day washout period and administration of the alternate formulation. Serial blood samples for pharmacokinetic assessment were collected at 0 hours (predose) up to 8 hours postdose. The plasma concentrations of capecitabine were analyzed by LC/MS-MS. Pharmacokinetic parameters (non-compartmental model) were assessed with WinNonlin software. The pharmacokinetic parameters assessed were area under the plasma concentration-time curve from time 0 to the time of last measurable concentration (AUC0-t), AUC from time zero to infinity (AUC0-∞), the peak plasma concentration of the drug (C max ), time needed to reach maximum concentration (Tmax), the elimination half-life (t1/2), and terminal elimination rate (λz). All were analyzed using an ANOVA model after logarithmic transformation of the data. For establishing bioequivalence (BE) for capecitabine， reference-scaled average bioequivalence (RSABE) acceptance criteria and average bioequivalence (ABE) acceptance criteria were used. Safety and tolerability was assessed during the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically conﬁrmed colorectal or breast cancer receiving capecitabine monotherapy or combination chemotherapy.
* Eligible patients were within 18-70 years of age.
* ECOG score was 0-2.
* Left ventricular ejection fraction (LVEF) > 50%.
* There was no serious persistent toxicity to capecitabine treatment before screening (laboratory tests ≤ grade 1 (NCI CTCAE 5.0 standard)
* Hand-foot syndrome ≤ grade 2 after recovery from the previous treatment period).

Exclusion Criteria:

* Patients were known allergy to fluorouracil or 5-fluorouracil.
* Patients with complete lack of known dihydropyrimidine dehydrogenase (DPD) activity.
* Patients with abnormal hepatic and renal function (serum creatinine≤ 1.5 ×ULN; CLcr ≥ 51 mL/min; bilirubin≤ 1.5 ×ULN; AST, ALT≤2.5×ULN)
* Needed to accept phenytoin, warfarin, other coumarin derivatives anticoagulants, folic acid, and CYP2C9 substrates during the research.
* Patients with brain metastases or other metastases of the central nervous system (except those who were treated at least 6 months prior to the start of the study and were stable and asymptomatic).

Ages: 28 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-26 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 18 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 18 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 18 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 18 days
  Adverse events were recorded to evaluate the safety of the studied drugs.

CONTACTS AND LOCATIONS:
Overall Officials: yu Cao, Doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase Ⅰ Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Qilu Pharmaceutical Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor.

REFERENCES:
- [Derived] Wang CJ, Li T, Lin PP, Tao Y, Jiang X, Li X, Wen Q, Cao Y. Pharmacokinetic and Safety Comparison of Two Capecitabine Tablets in Patients with Colorectal or Breast Cancer Under Fed Conditions: A Multicenter, Randomized, Open-Label, Three-Period, and Reference-Replicated Crossover Study. Adv Ther. 2021 Sep;38(9):4798-4814. doi: 10.1007/s12325-021-01817-4. Epub 2021 Aug 4. PMID 34347254